CLINICAL TRIAL: NCT00407823
Title: An Outcomes Comparison of ACCM/PALS Guidelines For Pediatric Septic Shock With and Without Central Venous Oxygen Saturation Monitoring
Brief Title: Comparison of Pediatric Septic Shock Treatment With and Without Central Venous Oxygen Saturation Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004/07949-7
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Child; Septic shock; Resuscitation; Central venous oxygen saturation; Cardiac output; Goal-directed therapy
MeSH Terms: conditions — Sepsis; Shock, Septic

INTERVENTIONS:
Procedure: Central venous oxygen saturation continuous monitoring

SUMMARY:
The purpose of this study was to compare ACCM/PALS guidelines performed with and without central venous oxygen saturation monitoring on the morbidity and mortality rate of children with severe sepsis and septic shock.

DETAILED DESCRIPTION:
Background: ACCM/PALS guidelines addresses early correction of pediatric septic shock using physical examination supplemented by indirect measures of cardiac output such as central venous or superior vena cava oxygen saturation (ScvO2>70%) in a goal directed approach. However, these endpoints are based on unsupported evidence. The purpose of this study was to compare ACCM/PALS guidelines performed with and without ScvO2 on the morbidity and mortality rate of children with severe sepsis and septic shock.

Methods: Children and adolescents with severe sepsis or fluid-refractory septic shock were recruited at two university-affiliated hospitals and randomly assigned to ACCM/PALS without, or with an ScvO2 goal directed (goal ScvO2 > 70%) resuscitation. Twenty-eight day mortality is the primary end point.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe sepsis or fluid-refractory septic shock that had not responded after 40 mL/kg of any resuscitation fluid or that required cardiovascular agents at any time during resuscitation

Exclusion Criteria:

* refusal to sign the written informed consent
* age less than 1 month or older than 19 years
* uncorrected cyanotic heart disease
* patients receiving exclusive palliative care
* patients that arrived from other hospitals more than 6 hours after the diagnosis of severe sepsis or septic shock.

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 268
Dates: Start 2004-01; Study Completion 2005-08

PRIMARY OUTCOMES:
28-day mortality

SECONDARY OUTCOMES:
Number of organ dysfunction
Administered treatments
Duration of cardiovascular agents therapy
Duration of mechanical ventilation
Length of Pediatric Intensive Care Unit stay
Days free of cardiovascular agents
Days free of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Claudio F Oliveira, MD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Instituto da Criança - HC-FMUSP, São Paulo, São Paulo
  - Hospital Universitário - USP, São Paulo, São Paulo

REFERENCES:
- [Result] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Derived] de Oliveira CF, de Oliveira DS, Gottschald AF, Moura JD, Costa GA, Ventura AC, Fernandes JC, Vaz FA, Carcillo JA, Rivers EP, Troster EJ. ACCM/PALS haemodynamic support guidelines for paediatric septic shock: an outcomes comparison with and without monitoring central venous oxygen saturation. Intensive Care Med. 2008 Jun;34(6):1065-75. doi: 10.1007/s00134-008-1085-9. Epub 2008 Mar 28. PMID 18369591